CLINICAL TRIAL: NCT00080951
Title: Phase II Trial Of Irinotecan + 5-Fluorouracil + Leucovorin + Oxaliplatin As First-Line Treatment For Metastatic Colorectal Cancer
Brief Title: Irinotecan, Fluorouracil, Leucovorin, and Oxaliplatin as First-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0341; NCI-2012-02581 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000357571 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- irinotecan + oxaliplatin + leucovorin + fluorouracil (Experimental): Patients receive irinotecan IV over 90 minutes and oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV and fluorouracil IV over 90 minutes on days 2-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline, before each chemotherapy course, and at the end of treatment.
  Patients are followed every 3 months until 5 years after registration.
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy as first-line therapy in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the tumor response rate in patients with metastatic colorectal cancer treated with irinotecan, fluorouracil, leucovorin calcium, and oxaliplatin as first-line treatment.

Secondary

* Determine the time to tumor progression, time to treatment failure, and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.
* Determine whether UGT1A1 polymorphism is related to toxicity (especially leukopenia, diarrhea, or neutropenia) or response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive irinotecan IV over 90 minutes and oxaliplatin IV over 2 hours on day 1 and leucovorin calcium IV and fluorouracil IV over 90 minutes on days 2-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each chemotherapy course, and at the end of treatment.

Patients are followed every 3 months until 5 years after registration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma

  * Metastatic disease
* Not curable by surgery or amenable to radiotherapy with curative intent
* Measurable disease

  * Patients with only lesions measuring ≥ 1 cm but < 2 cm must use spiral CT scan for pre- and post-treatment tumor assessments
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST ≤ 5 times upper limit of normal (ULN)
* Bilirubin ≤ 0.5 mg/dL above ULN

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No unstable angina
* No symptomatic congestive heart failure
* No serious uncontrolled cardiac arrhythmia

Pulmonary

* No prior clinical diagnosis of interstitial lung disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or uncontrolled infection
* No other concurrent serious illness
* No pre-existing paraesthesias/dysesthesias of ≥ grade 2 that would interfere with function
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinomas

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent sargramostim (GM-CSF)

Chemotherapy

* At least 6 months since prior adjuvant chemotherapy
* No prior fluorouracil for advanced colorectal cancer
* No prior adjuvant oxaliplatin
* No prior adjuvant irinotecan

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to > 25% of bone marrow

Surgery

* At least 4 weeks since prior major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-03; Primary Completion 2005-04 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
tumor response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
overall survival | Up to 5 years
time to treatment failure | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] McWilliams RR, Goetz MP, Morlan BW, Salim M, Rowland KM, Krook JE, Ames MM, Erlichman C. Phase II trial of oxaliplatin/irinotecan/5-fluorouracil/leucovorin for metastatic colorectal cancer. Clin Colorectal Cancer. 2007 May;6(7):516-21. doi: 10.3816/CCC.2007.n.017. PMID 17553200